CLINICAL TRIAL: NCT03241238
Title: The Effect of Dietary Fiber on Food Liking
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: No effect was found
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Faculty Advisor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UTK IRB-17-03817-XP
Record Dates: First submitted 2017-07-25; First posted 2017-08-07 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Different Fermentable Fiber; Satiation
MeSH Terms: interventions — Eating

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Regular Brownie (Other): Regular Brownie For the regular brownie condition (RB), participants will consume the brownie preload and then consume a meal 20 minutes later.
  Interventions: Other: Eating
- Psyllium Brownie (Other): For the psyllium brownie (PG), participants will consume a psyllium brownie and then consume a meal 20 minutes later.
  Interventions: Other: Eating
- β-glucan Brownie (Other): For the β-glucan Brownie (BG), participants will consume a β-glucan Brownie preload and then consume a meal 20 minutes later
  Interventions: Other: Eating

INTERVENTIONS:
Other: Eating — Participants will have 10 minutes to eat all of the brownie and drink 6 oz of water. They will then have 20 minutes to eat as much or as little of a meal (consisting of a sandwich, grapes and chips).

SUMMARY:
This study will investigate the effects of different fermenting fibers on liking of foods.

DETAILED DESCRIPTION:
Participants will be randomized to one of three orders to reduce the possibility of an order effect.The participants will be given a brownie specific for the condition they are in and then will be instructed to eat the brownie in 10 minutes. Twenty minutes after consuming the brownie participants will be served a lunch. Dependent variables will be food liking.

At the start of the session the participant will be asked to recall all foods and beverages consumed 24 hours prior to the scheduled appointment. During this recall if a participant reports consuming any foods or beverages besides water within 3 hours of the appointment, the appointment will be rescheduled. Participants will also be asked if they have participated in any physical activity 24 hours prior to their scheduled appointment. If the participant answers "yes," then the appointment will be rescheduled.

After completing hunger and fullness VAS, participants will be presented with a preload of brownie, β-glucan brownie, or psyllium brownie. The brownie will be prepared from the same base recipe, thus be of the same approximate energy and macronutrient composition, but differ in amount and type of dietary fiber. The base recipe will use a box of Pillsbury™ dark chocolate brownie mix, two eggs, ¼ cup water and 2/3 cup of Food Club™ unsweetened applesauce. The regular brownie will not contain any fiber, while the β-glucan and psyllium brownie will contain about 6 grams of their respective fiber: Bulk Supplements™ β-glucan and Frontier™ Psyllium Husk Powder. An additional tablespoon of water will be added to the β-glucan brownie mix. The brownie will be presented warm, with two tablespoons of Cool Whip™ fat free spread on top, with 6 ounces of water. The participants will be told to consume all of the brownie and toping, and to drink all of the 6 oz of water within 10 minutes. Next, participants will rate their hunger and fullness again with the VAS and sit quietly for 20 minutes reading current magazines (i.e., People, Entertainment Weekly). After 20 minutes, the participants will be presented with a sandwich (turkey or ham), chips, and grapes.The sandwich will be cut into quarters on a plate, the chips and grapes will be presented in two separate bowls. Following the presentation of the meal, participants will be instructed that they will have 20 minutes to eat as much or as little as they would like of the meal provided until satisfied, however they need to at least taste each of the foods. At the completion of 20 minutes, the lunch will be removed and the participant will be asked to complete a scale for evaluating levels of hunger, fullness, and liking of the foods.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 to 24.9 kg/m^2
* Unrestrained eater (<12 on Three Factor Eating Questionnaire [TFEQ])
* report liking turkey or ham sandwiches, brownies, grapes, and potato chips (rate all items >50mm on a visual analogue scale [VAS]).
* Report regularly eating before 10 am
* Can completed all sessions within 6 weeks of the screening session.

Exclusion Criteria:

* Report binge eating
* Report a medical condition that influences eating
* Report food allergies to the study foods
* Currently smoke
* Report dietary restrictions
* Report not liking brownies
* Report currently taking a medication that effects appetite
* Report being pregnant or breast-feeding
* Report being an athlete in training.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Hunger | Change across the meal, 20 minutes
  100 mm Visual analog scale
Fullness | Change across the meal, 20 minutes
  100 mm Visual analog scale
Liking | Change across the meal, 20 minutes
  100 mm Visual analog scale

CONTACTS AND LOCATIONS:
Locations (1):
- Healthy Eating and Activity Laboratory, University of Tennessee, Knoxville, Tennessee, United States

REFERENCES:
- [Background] Raynor HA, Epstein LH. Effects of sensory stimulation and post-ingestive consequences on satiation. Physiol Behav. 2000 Sep 15;70(5):465-70. doi: 10.1016/s0031-9384(00)00291-2. PMID 11110999
- [Background] Rebello CJ, O'Neil CE, Greenway FL. Dietary fiber and satiety: the effects of oats on satiety. Nutr Rev. 2016 Feb;74(2):131-47. doi: 10.1093/nutrit/nuv063. Epub 2016 Jan 2. PMID 26724486
- [Background] Brum JM, Gibb RD, Peters JC, Mattes RD. Satiety effects of psyllium in healthy volunteers. Appetite. 2016 Oct 1;105:27-36. doi: 10.1016/j.appet.2016.04.041. Epub 2016 May 7. PMID 27166077
- [Background] Delargy HJ, O'Sullivan KR, Fletcher RJ, Blundell JE. Effects of amount and type of dietary fibre (soluble and insoluble) on short-term control of appetite. Int J Food Sci Nutr. 1997 Jan;48(1):67-77. doi: 10.3109/09637489709006965. PMID 9093551
- [Background] McRorie JW Jr, McKeown NM. Understanding the Physics of Functional Fibers in the Gastrointestinal Tract: An Evidence-Based Approach to Resolving Enduring Misconceptions about Insoluble and Soluble Fiber. J Acad Nutr Diet. 2017 Feb;117(2):251-264. doi: 10.1016/j.jand.2016.09.021. Epub 2016 Nov 15. PMID 27863994
- [Background] Ridgway PS, Jeffrey DB. A comparison of the Three-Factor Eating Questionnaire and the Restraint Scale and consideration of Lowe's Three-Factor Model. Addict Behav. 1998 Jan-Feb;23(1):115-8. doi: 10.1016/s0306-4603(97)00031-2. PMID 9468749
- [Background] Stunkard AJ, Messick S. The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. J Psychosom Res. 1985;29(1):71-83. doi: 10.1016/0022-3999(85)90010-8. PMID 3981480
- [Background] Lohman TR, Roche AF, Martorell R. Anthropometric Standardization Reference Manual. Champaign,Illinois: Human Kinetics Books; 1988.
- [Background] Overweight and Obesity Statistics. (2012). Retrieved February 10, 2017, from https://www.niddk.nih.gov/health-information/health-statistics/Pages/overweight-obesity-statistics.aspx